CLINICAL TRIAL: NCT00577525
Title: Viral Infection of Lymphoid Cells Occuring at the First Manifestation of Idiopathic Nephrotic Syndrome
Brief Title: Latent Viral Infection of Lymphoid Cells in Idiopathic Nephrotic Syndrome
Acronym: Nephrovir
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P070126
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: NEPHROSIS, LIPOID
Keywords: LATENT VIRAL INFECTION; GENOME HYBRIDIZATION; HERPES VIRUS; ADENOVIRUS
MeSH Terms: conditions — Nephrosis, Lipoid; Adenoviridae Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, red cells and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Case : Patients with steroid sensitive nephrotic syndrome
- 2: Controls (matched for age and sexe with the first group)

SUMMARY:
The primary purpose of the study is to evaluate the association of a latent infection of lymphoid cells during the first manifestation of steroid sensitive nephrite syndrome. The thirty nine units of general pediatrics and pediatric nephrite covering the parisian area will participate to the study. We speculate that hybridization of the genome, or a part of the genome, of a virus in lymphoid cells is responsible specific changes of genes expression, leading to the development of the disease.

DETAILED DESCRIPTION:
An additional blood volume will be sampled in patients and controls during a scheduled biological check-up for the initial disease and viral genome of EBV, CMV, HHV6, HHV7 as well as adenovirus will be searched for using PCR reaction in total blood DNA extract. The frequency of a latent hybridization of virus genome within human genome will be compared between patients with steroid sensitive nephrotic syndrome and controls matched for age and sex. Secondary studies will include a comparison of steroid dependency in nephrotic patients according to the occurence of a latent viral hybridization, the epidemiology of idiopathic nephrotic syndrome in the Parisian area and a pharmacogenetic analysis of steroid sensitivity and dependency. If necessary, the chromosomal localization of viral hybridization will be studied with fluorescence in situ hybridization using specific probes.

ELIGIBILITY:
Inclusion Criteria:

* proteinuria over 0.25 g/mmol of creatinine with hypoalbuminemia below 30g/L for the case
* No history of renal disease
* Normal C3 and negativity for hepatitis B and C

Exclusion Criteria:

* no medical insurance
* inclusion in another study

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From the thirty nine units of general pediatrics and pediatric nephrology covering the Parisian area
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Hybridization of viral genome will be studied at the first manifestation of idiopathic nephrotic syndrome | Within the 3 days of the first manifestation

SECONDARY OUTCOMES:
Steroid sensitivity will be checked by 1 month of prednisone therapy according to the recommendation of the " SOCIETE DE NEPROLOGIE PEDIATRIQUE" and steroid dependency will be checked at 4.5 months of prednisone therapy. | 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Georges DESCHENES, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Robert Debre, Paris, France

REFERENCES:
- [Result] Sellier-Leclerc AL, Duval A, Riveron S, Macher MA, Deschenes G, Loirat C, Verpont MC, Peuchmaur M, Ronco P, Monteiro RC, Haddad E. A humanized mouse model of idiopathic nephrotic syndrome suggests a pathogenic role for immature cells. J Am Soc Nephrol. 2007 Oct;18(10):2732-9. doi: 10.1681/ASN.2006121346. Epub 2007 Sep 12. PMID 17855645
- [Result] Ulinski T, Perrin L, Guigonis V, Driss F, Deschenes G, Bensman A. Remission of steroid- and CyA-resistant nephrotic syndrome using multiple drug immunosuppression. Pediatr Nephrol. 2007 Oct;22(10):1723-6. doi: 10.1007/s00467-007-0551-x. Epub 2007 Jul 17. PMID 17636340
- [Result] Doucet A, Favre G, Deschenes G. Molecular mechanism of edema formation in nephrotic syndrome: therapeutic implications. Pediatr Nephrol. 2007 Dec;22(12):1983-90. doi: 10.1007/s00467-007-0521-3. Epub 2007 Jun 7. PMID 17554565
- [Result] Lorton F, Raynot J, Letavernier B, Isapof A, Debiec H, Pressac M, Deschenes G, Lenoir M, Ross-Cerdan L, Grapin C, Bensman A, Ulinski T. Gross proteinuria post transplant in a child with nephrotic syndrome of the Finnish type--mechanical vs immunological pathogenesis. Nephrol Dial Transplant. 2006 Dec;21(12):3579-82. doi: 10.1093/ndt/gfl459. Epub 2006 Aug 25. No abstract available. PMID 16935903
- [Result] Lourdel S, Loffing J, Favre G, Paulais M, Nissant A, Fakitsas P, Creminon C, Feraille E, Verrey F, Teulon J, Doucet A, Deschenes G. Hyperaldosteronemia and activation of the epithelial sodium channel are not required for sodium retention in puromycin-induced nephrosis. J Am Soc Nephrol. 2005 Dec;16(12):3642-50. doi: 10.1681/ASN.2005040363. Epub 2005 Nov 2. PMID 16267158
- [Result] Nathanson S, Cochat P, Andre JL, Guyot C, Loirat C, Nivet H, Deschenes G. Recurrence of nephrotic syndrome after renal transplantation: influence of increased immunosuppression. Pediatr Nephrol. 2005 Dec;20(12):1801-4. doi: 10.1007/s00467-005-2053-z. Epub 2005 Oct 14. PMID 16228184
- [Result] Mansour H, Cheval L, Elalouf JM, Aude JC, Alyanakian MA, Mougenot B, Doucet A, Deschenes G. T-cell transcriptome analysis points up a thymic disorder in idiopathic nephrotic syndrome. Kidney Int. 2005 Jun;67(6):2168-77. doi: 10.1111/j.1523-1755.2005.00322.x. PMID 15882260
- [Result] Frange P, Frey MA, Deschenes G. [Immunity and immunosuppression in childhood idiopathic nephrotic syndrome]. Arch Pediatr. 2005 Mar;12(3):305-15. doi: 10.1016/j.arcped.2004.12.015. French. PMID 15734130
- [Result] Deschenes G, Feraille E, Doucet A. [Cellular and molecular mechanisms of sodium pump activation in experimental models of nephrotic syndrome]. Nephrologie. 2003;24(3):121-6. French. PMID 12814058
- [Result] Feraille E, Mordasini D, Gonin S, Deschenes G, Vinciguerra M, Doucet A, Vandewalle A, Summa V, Verrey F, Martin PY. Mechanism of control of Na,K-ATPase in principal cells of the mammalian collecting duct. Ann N Y Acad Sci. 2003 Apr;986:570-8. doi: 10.1111/j.1749-6632.2003.tb07255.x. PMID 12763891
- [Result] Debiec H, Guigonis V, Mougenot B, Haymann JP, Bensman A, Deschenes G, Ronco PM. Antenatal membranous glomerulonephritis with vascular injury induced by anti-neutral endopeptidase antibodies: toward new concepts in the pathogenesis of glomerular diseases. J Am Soc Nephrol. 2003 Jun;14 Suppl 1:S27-32. doi: 10.1097/01.asn.0000067649.64849.75. No abstract available. PMID 12761235
- [Result] Deschenes G, Feraille E, Doucet A. Mechanisms of oedema in nephrotic syndrome: old theories and new ideas. Nephrol Dial Transplant. 2003 Mar;18(3):454-6. doi: 10.1093/ndt/18.3.454. No abstract available. PMID 12584259
- [Result] Nathanson S, Lucidarme N, Landman-Parker J, Deschenes G. Long-term survival of renal graft complicated with Burkitt lymphoma. Pediatr Nephrol. 2002 Dec;17(12):1066-8. doi: 10.1007/s00467-002-0992-1. Epub 2002 Oct 8. PMID 12478360
- [Result] Deschenes G. [LMXb1 generates the morphology of podocytes]. Arch Pediatr. 2002 Sep;9(9):1002-3. doi: 10.1016/s0929-693x(02)00071-4. No abstract available. French. PMID 12387184